CLINICAL TRIAL: NCT01560104
Title: Randomized, Double-Blind, Multicenter, Phase 2 Trial Comparing Veliparib Plus Carboplatin and Paclitaxel Versus Placebo Plus Carboplatin and Paclitaxel in Previously Untreated Metastatic or Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Clinical Study Conducted in Multiple Centers Comparing Veliparib in Combination With Carboplatin and Paclitaxel Versus a Placebo in Combination With Carboplatin and Paclitaxel in Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-898; 2011-003427-36 (EudraCT Number)
Record Dates: First submitted 2012-02-29; First posted 2012-03-22 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Non-Small -Cell Lung Cancer
Keywords: Randomized; metastatic; ABT-888; paclitaxel; non-small cell lung cancer; PARP; veliparib; progression free survival; carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — veliparib; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- veliparib and carboplatin and paclitaxel (Experimental): Veliparib on Days 1-7 and carboplatin and paclitaxel on Day 3 of a 21 day cycle
  Interventions: Drug: Veliparib; Drug: Carboplatin; Drug: paclitaxel
- placebo and carboplatin and paclitaxel (Placebo Comparator): Placebo on Days 1-7 and carboplatin and paclitaxel on Day 3 of a 21 day cycle
  Interventions: Drug: Carboplatin; Drug: paclitaxel; Drug: placebo

INTERVENTIONS:
Drug: Veliparib
  Other Names: ABT-888
  Arms: veliparib and carboplatin and paclitaxel
Drug: Carboplatin
Drug: paclitaxel
Drug: placebo
  Arms: placebo and carboplatin and paclitaxel

SUMMARY:
A Randomized, Double-Blind, Multicenter, Phase 2 Trial Comparing Veliparib Plus Carboplatin and Paclitaxel Versus Placebo Plus Carboplatin and Paclitaxel in Previously Untreated Metastatic or Advanced Non-Small-Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Subjects will be randomized in a 2:1 ratio to one of the two treatment groups. The safety of each treatment group will be assessed by evaluating study drug exposure, adverse events, serious adverse events, all deaths, changes in laboratory determinations and vital sign parameters. Progression -Free Survival (PFS) using Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1) will be assessed as well as Overall Survival (OS) and the Objective Response Rate (ORR). Study visits will be conducted according to the protocol schedule. Study visits will include physical examination, laboratory blood sample collection, and assessment of vital signs, medical history and urinalysis. 12-lead Electrocardiogram (ECG) will be performed at protocol specified visits.

ELIGIBILITY:
Inclusion Criteria: - Life expectancy > 12 weeks (as per Investigator's clinical assessment).

* Subject must have cytologically or histologically confirmed non-small cell lung cancer (NSCLC).
* Subject must have metastatic or advanced non-small cell lung cancer (NSCLC) (stage IIIB or IV) that is not amenable to surgical resection or radiation with curative intent at time of study Screening.
* Subject must have at least 1 unidimensional measurable non-small cell lung cancer (NSCLC) lesion on a Computed Tomography (CT) scan as defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1).
* Subject must consent to provide available archived formalin fixed, paraffin embedded (FFPE) tissue sample of non-small cell lung cancer (NSCLC) lesion (primary or metastatic) for central review and biomarker analysis.
* Subject must have no history of brain metastases or evidence of primary central nervous system (CNS) tumors as demonstrated by a baseline magnetic resonance imaging (MRI).
* Subject must have an Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1.
* Subjects with fluid retention, including ascites or pleural effusion, may be allowed at the discretion of the Investigator.

Exclusion Criteria: -Subject has a known hypersensitivity to paclitaxel or to other drugs formulated with polyethoxylated castor oil (Cremophor).

* Subject has a known hypersensitivity to platinum compounds.
* Subjects with peripheral neuropathy ≥ grade 2.
* Subjects with a known epidermal growth factor receptor (EGFR) mutation of exon 19 deletion or L858R mutation in exon 21. (Subjects with wild type epidermal growth factor receptor (EGFR), unknown status or other type of epidermal growth factor receptor (EGFR) mutation will be considered eligible).
* Subject has received prior systemic anti-cancer therapy for metastatic non-small cell lung cancer (NSCLC).
* Subject has received adjuvant chemotherapy ≤ 12 months prior to Cycle 1 Day 1.
* Subject has received anti-cancer Chinese medicine or anti-cancer herbal remedies within 14 days prior to Cycle 1 Day 1.
* Subject has undergone External Beam Radiation Therapy (EBRT) ≤ 8 weeks prior to Cycle 1 Day 1.
* Clinically significant and uncontrolled major medical condition(s).
* Subject has previously been treated with a poly-(ADP-ribose)-polymerase (PARP) inhibitor

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Radiographic evaluation starting from the third day of study treatment and on average every 6 weeks until documented progression or date of death from any cause, whichever came first, until patient is registered as off study.

SECONDARY OUTCOMES:
Overall Survival (OS) | Monthly after patient is registered off study up to 36 months or until date of death from any cause, whichever came first.
  Continuously from date of randomization until date of death from any cause or until patient is registered as off study, whichever came first.
Objective Response Rate (ORR) | Radiographic evaluation starting from the third day of study treatment and on average every 6 weeks until documented progression or date of death from any cause, whichever came first, until patient is registered as off study.
Chemotherapy Induced Peripheral Neuropathy (CIPN) | From date of screening, first day of study treatment and then every cycle (about every 3 weeks) until date of death from any cause or patient is registered as off study, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Giranda, MD, Study Director — AbbVie

REFERENCES:
- [Derived] Ramalingam SS, Blais N, Mazieres J, Reck M, Jones CM, Juhasz E, Urban L, Orlov S, Barlesi F, Kio E, Keiholz U, Qin Q, Qian J, Nickner C, Dziubinski J, Xiong H, Ansell P, McKee M, Giranda V, Gorbunova V. Randomized, Placebo-Controlled, Phase II Study of Veliparib in Combination with Carboplatin and Paclitaxel for Advanced/Metastatic Non-Small Cell Lung Cancer. Clin Cancer Res. 2017 Apr 15;23(8):1937-1944. doi: 10.1158/1078-0432.CCR-15-3069. Epub 2016 Oct 10. PMID 27803064